CLINICAL TRIAL: NCT01354990
Title: Sitagliptin (JANUVIA®) Post Marketing Surveillance Protocol
Brief Title: A Post Marketing Safety Study of Sitagliptin (JANUVIA®) (MK-0431-234)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0431-234
Record Dates: First submitted 2011-05-16; First posted 2011-05-17 (Estimated); Results first posted 2012-06-04 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants treated with sitagliptin
  Interventions: Drug: Sitagliptin (JANUVIA®)

INTERVENTIONS:
Drug: Sitagliptin (JANUVIA®) — Participants prescribed Sitagliptin (JANUVIA®) in routine clinical practice.

SUMMARY:
The primary objective of this study is to obtain safety information on the use of sitagliptin (JANUVIA®) from endocrinologists, diabetologists, internists, and general practitioners.

ELIGIBILITY:
Inclusion Criteria:

- Must be taking sitagliptin (JANUVIA™) for the treatment of type 2 diabetes

mellitus

- Treating physician must agree to provide information regarding the participants treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with type 2 diabetes mellitus who are treated with sitagliptin as per the standard of care in a physician's practice
Sampling Method: Non-Probability Sample
Enrollment: 2974 (Actual)
Dates: Start 2009-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a postmarketing, safety study of participants with Type 2 diabetes mellitus prescribed sitagliptin phosphate (JUNUVIA®) in clinical practices in the Philippines.
Groups:
- Sitagliptin Phosphate (JANUVIA®): Participants prescribed Sitagliptin Phosphate (JANUVIA®) in routine clinical practice.
Period: Overall Study
Arm/Group | Sitagliptin Phosphate (JANUVIA®)
Started | 2974
Completed | 2974
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sitagliptin Phosphate (JANUVIA®)
Number analyzed (Participants) | 2974
Age, Customized [Number; unit: participants]
  0 - 19 | 0 (12.2)
  20 - 99 | 2926
  Unspecified | 48
Sex/Gender, Customized [Number; unit: participants]
  Female | 1577
  Male | 1351
  Unspecified | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Adverse Event
Time Frame: Up to approximately 28 months
Measure: Number; unit: participants
Arm/Group | Sitagliptin Phosphate (JANUVIA®)
Number analyzed (Participants) | 2974
participants | 25

2. Primary Outcome: Age of Participants Prescribed Sitagliptin
Time Frame: Up to approximately 28 months
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Sitagliptin Phosphate (JANUVIA®)
Number analyzed (Participants) | 2974
years | 55 (12.2)

3. Primary Outcome: Number of Participants With Concomitant Therapies
Time Frame: Up to approximately 28 months
Measure: Number; unit: participants
Arm/Group | Sitagliptin Phosphate (JANUVIA®)
Number analyzed (Participants) | 2974
participants | 1878

4. Primary Outcome: Number of Participants With Concomitant Conditions
Time Frame: Up to approximately 28 months
Measure: Number; unit: participants
Arm/Group | Sitagliptin Phosphate (JANUVIA®)
Number analyzed (Participants) | 2974
participants | 752

ADVERSE EVENTS:
Time Frame: Up to approximately 28 months
Arm/Group | Sitagliptin Phosphate (JANUVIA®)
Serious Adverse Events (participants affected / at risk) | 0/2974
Other Adverse Events (participants affected / at risk) | 0/2974

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No